CLINICAL TRIAL: NCT06372353
Title: The Effect Of Baduanjin Exercises On Functional Capacity, Respiratory Functions And Quality Of Life In Patients With Idiopathic Pulmonary Fibrosis: a Randomized Controlled Study
Brief Title: The Effect Of Baduanjin Exercises In Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 777
Record Dates: First submitted 2024-03-13; First posted 2024-04-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Fibrosis, Idiopathic
Keywords: Idiopathic Pulmonary Fibrosis; Baduanjin Exercise; Functional Capacity; Respiratory Function Tests; Quality of Life
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention Group (Experimental): The subjects in the intervention group were given 24 sessions of supervised online Baduanjin exercise training
  Interventions: Other: Baduanjin Exercise
- Control Group (No Intervention)

INTERVENTIONS:
Other: Baduanjin Exercise — Baduanjin exercise training program was applied to the subjects in the exercise group, 3 days a week, 5 minutes each with warm-up and cool-down exercises, for a total of 24 sessions, 60 minutes each, under supervision, online, via the ZOOM application, for 8 weeks. In addition, the patients did the exercises unsupervised at home once a week. The patients' first sessions were held in the hospital
  Other Names: exercise
  Arms: intervention Group

SUMMARY:
Introduction and Objectives:IPF, characterized by shortness of breath and progressive deterioration in lung function.Baduanjin (BJ) is a mindbody health exercise that combines physical exercise with psychological properties to maximize both physical and mental health.The aim of the study is to investigate the effectiveness of these exercises in patients with IPF and to present an alternative in terms of the applicability of BJ exercises as a new treatment method

Methods: 28 volunteers were invited to the study.These patients were randomly divided into 2 groups.The subjects in the exercise group were given 24 sessions of supervised online BJ exercise training, 3 days a week, for 8 weeks. The patients included in the control group did not receive any training during the 8 week period

DETAILED DESCRIPTION:
Introduction and Objectives: Idiopathic Pulmonary Fibrosis (IPF) is a disease with a poor prognosis that causes fibrosis in the interstitial space of the lungs, characterized by shortness of breath and progressive deterioration in lung function. The main purpose of this randomized controlled study is to investigate the effectiveness of applying Baduanjin exercise training for 8 weeks, which has previously been shown to be effective in other patient groups, on respiratory functions (%FVC, FEV1, FEV1%), respiratory muscle strength (MIP and MEP) and quality of life (SGRQ) in patients with IPF. It is planned to be used as a new treatment method in this patient group. It is to offer an alternative in terms of the applicability of Baduanjin exercises.

Methods: Twenty eight volunteers were invited to the study. These patients were randomly divided into 2 groups. The subjects in the exercise group were given 24 sessions of supervised online Baduanjin exercise training, 3 days a week for 8 weeks, and the patients also did Baduanjin exercise 1 day a week at home unattended. The first evaluation, follow-up and final evaluation of the patients included in the control group were performed; In addition to their sociodemographic characteristics, functional exercise capacity, respiratory muscle strength and respiratory functions, quality of life were evaluated before and after treatment.

Keywords: Idiopathic Pulmonary Fibrosis, Baduanjin exercise, Functional capacity, Respiratory functions, Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with IPF according to international guideline criteria; Medical Research Council (mMRC) dyspnea score < 5; being able to ambulate without using an assistive device; being between the ages of 18-75; being cooperative; a stable patient with no pulmonary exacerbation in the last 6 weeks; having no vision or hearing deficits; having the necessary internet and computer or telephone equipment to participate in the online exercise program.

Exclusion Criteria:

* Participation in a formal rehabilitation program no later than 4 months before the beginning of the study; having severe musculoskeletal or neurological disorders; having severe heart disease; inability to understand informed consent conditions and exercises; need for additional oxygen at rest; presence of obvious lung infection requiring anti-infection therapy (patients had a respiratory tract infection or systemic infection within 4 weeks before enrollment); situations where exercise is contraindicated; presence of another chronic lung disease (e.g., collagen vascular disease, obstructive pulmonary disease, nonparenchymal restrictive lung disease, occupational lung disease, sarcoidosis, or other idiopathic interstitial pneumonia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Functional capacity | Baseline of the study and 8 weeks after intervention
  Functional exercise capacity was evaluated with the six-minute walking test (6MWT). Participants rested in a sitting position for 10 minutes before starting the test. Participants were then explained the test protocol and asked to walk as far as possible without running in a 30-meter straight corridor for six minutes. At the end of the test, the evaluations made before the test were repeated and the six-minute walking distance (6MWD) was recorded in meters

SECONDARY OUTCOMES:
Pulmonary Function Tests | Baseline of the study and 8 weeks after intervention
  Pulmonary function tests were performed using standard references. Portable spirometry (Spirobank II; MIR, Rome, Italy) was utilized to assess pulmonary functions. The assessments adhered to the standards outlined by the American Thoracic Society (ATS) and the European Respiratory Society (ERS) guidelines, with measurements expressed as percentages of predicted values. The following parameters related to pulmonary function were measured: Forced expiratory volume in 1 second (FEV1).
Pulmonary Function Tests | Baseline of the study and 8 weeks after intervention
  Pulmonary function tests were performed using standard references. Portable spirometry (Spirobank II; MIR, Rome, Italy) was utilized to assess pulmonary functions. The assessments adhered to the standards outlined by the American Thoracic Society (ATS) and the European Respiratory Society (ERS) guidelines, with measurements expressed as percentages of predicted values. The following parameters related to pulmonary function were measured: Forced vital capacity (FVC).
Pulmonary Function Tests | Baseline of the study and 8 weeks after intervention
  Pulmonary function tests were performed using standard references. Portable spirometry (Spirobank II; MIR, Rome, Italy) was utilized to assess pulmonary functions. The assessments adhered to the standards outlined by the American Thoracic Society (ATS) and the European Respiratory Society (ERS) guidelines, with measurements expressed as percentages of predicted values. The following parameters related to pulmonary function were measured: Peak expiratory flow (PEF).
Pulmonary Function Tests | Baseline of the study and 8 weeks after intervention
  Pulmonary function tests were performed using standard references. Portable spirometry (Spirobank II; MIR, Rome, Italy) was utilized to assess pulmonary functions. The assessments adhered to the standards outlined by the American Thoracic Society (ATS) and the European Respiratory Society (ERS) guidelines, with measurements expressed as percentages of predicted values. The following parameters related to pulmonary function were measured: Forced mid-expiratory flow (FEF).
Respiratory muscle strength | Baseline of the study and 8 weeks after intervention
  Respiratory muscle strengths (intraoral pressure measurement) were performed using standard references. Maximal inspiratory pressures (MIP) were utilized to assess the strength of the respiratory muscles. Participants; MIP were measured and documented according to ATS/ERS criteria using a portable MicroRPM device (Micro Medical, Basingstoke, UK) . The highest of the at least three measurements exhibiting a difference between them of no more than 5 cm H2O is documented for MIP. Determination of predicted value for MIP was made according to the definitions put forward by Black and Hyatt.
Respiratory muscle strength | Baseline of the study and 8 weeks after intervention
  Respiratory muscle strengths (intraoral pressure measurement) were performed using standard references. Maximal expiratory pressures (MEP) were utilized to assess the strength of the respiratory muscles. Participants; MEP were measured and documented according to ATS/ERS criteria using a portable MicroRPM device (Micro Medical, Basingstoke, UK) . The highest of the at least three measurements exhibiting a difference between them of no more than 5 cm H2O is documented for MEP. Determination of predicted value for MEP was made according to the definitions put forward by Black and Hyatt.
St. George's Respiratory Questionnaire | Baseline of the study and 8 weeks after intervention
  Quality of life was measured with using Saint George Respiratory Questionaire (SGRQ), SGRQ, a 76-question form which includes dimensions for SGRQ activity, SGRQ impact, SGRQ symptoms, and SGRQ total. Scale (score 0-100, where 100 is the worst). All assessments were performed for the same patient at similar times of the day.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University - Cerrahpaşa, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056